CLINICAL TRIAL: NCT05041790
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase IV Trial to Evaluate the Efficacy and Safety of Choline Alfoscerate Compared to Placebo in Patients With Degenerative Mild Cognitive Impairment(ESCALADE)
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Choline Alfoscerate Compared to Placebo in Patients With Degenerative Mild Cognitive Impairment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Choline Alfoscerate Re-evaluation Consortium (57 pharmaceutical companies) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B78_02MCI2003
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Choline Alfoscerate
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline Alfoscerate (Experimental)
  Interventions: Drug: Choline Alfoscerate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Choline Alfoscerate — Choline Alfoscerate 400mg per oral 3 times a day during the entire treatment period.
  Arms: Choline Alfoscerate
Drug: Placebo — Placebo of Choline Alfoscerate 400mg per oral 3 times a day during the entire treatment period.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, Phase IV trial to evaluate the efficacy and safety of Choline Alfoscerate compared to placebo in patients with degenerative mild cognitive impairment.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either Choline Alfoscerate or its placebo. Investigational Products(IP, Choline Alfoscerate or its placebo) will be administered 3 times a day per oral during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 55 years
2. Diagnosis of mild cognitive impairment due to Alzheimer's disease that meets NIA-AA criteria
3. Diagnosed with mild cognitive impairment on SNSB
4. Delayed recall score of SVLT ≤ "average -1.5 standard deviation"
5. K-MMSE-2 score ≥ 24
6. The CDR score 0.5, and the memory item score 0.5 or 1 point
7. Patients with caregivers who are in regular contact, can visit together
8. Walk or move using walking aids (i.e., walkers, walking sticks or wheelchairs)
9. Sufficient vision, hearing, language skills, motor skills, and understanding to follow the examination procedure.
10. Written informed consent

Exclusion Criteria:

1. Diagnosis of dementia (including secondary dementia due to Alzheimer's disease, vascular dementia, infections of the central nervous system (e.g., HIV, syphilis, Creutzfeld-Jacob disease), Pixie disease, Huntington's disease, Parkinson's disease, etc.)
2. Medication of dementia within the past three months
3. Brain functional improvement medication in the past six weeks.
4. Medication that may affect cognitive function during clinical trials
5. No studies (no regular school entrance), illiteracy
6. Significant neurological conditions (such as stroke, multiple sclerosis, severe head trauma with loss of consciousness, cerebral palsy, cerebral tumor, cerebral infarction, spinal infarction or central nervous system infection) and/or evidence (CT or MRI results performed within the past 12 months or during screening)
7. Abnormal results from Vitamin B12, Thyroid Stimulated Hormone Test (TSH), HIV-Ab, and VDRL test contribute to or contribute to cognitive impairment of the subject
8. Serious mental disorders such as severe depression, schizophrenia, alcoholism, drug dependence, etc.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects whose cognitive function is maintained/improved at 48 weeks compared to baseline | Baseline to 48 weeks
  Definition of maintained/improved of cognitive function: decreased by more than or equal to 0 point of modified ADAS-Cog score

SECONDARY OUTCOMES:
The proportion of subjects reduced by more than or equal to 0 points for modified ADAS-Cog score at 24 weeks compared to baseline | Baseline to 24 weeks
The proportion of subjects reduced by more than 2 points of modified ADAS-Cog score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
The proportion of subjects reduced by more than 4 points of modified ADAS-Cog score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
The change of Modified ADAS-Cog score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
  The Modified ADAS-Cog 13 scale has a total of 85 points, and the higher the score, the higher the severity.
The proportion of subjects increased by more than or equal to 0 point of K-MMSE-2 score at 24 and 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
The change of K-MMSE-2 score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
  K-MMSE-2 scale has a total of 30 points, and the lower the score, the higher the severity.
The change of CDR-SB score at 48 weeks compared to baseline | Baseline to 48 weeks
  CDR-SB calculates the CDR score as Sum of Boxes, in which case, the score in the six areas obtained by the evaluation is added as it is, and the range of the total score is 0 to 30, and the higher the score, the more severe the degree of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: JaeHong Lee, MD, Principal Investigator — Asan Medical Center Institutional Review Board
Locations (1):
- Asan Medical Center Institutional Review Board, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No